CLINICAL TRIAL: NCT06824441
Title: Symptom Reporting by Children, Adolescents and Young Adults With Cancer and Their Caregivers During a Clinic Visit: A Feasibility, Usability and Acceptability Study
Brief Title: Feasibility Usability & Acceptability Study: Symptom Reporting by Children Adolescents & Young Adults w/Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB- 71098; NCI-2025-00233 (Other: CTRP)
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Adolescent Behavior; Pediatric Cancer; Oncology
MeSH Terms: conditions — Adolescent Behavior; Neoplasms | interventions — Aging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ped-PRO-CTCAE Questionnaire Completion for Children, AYAs, Caregivers, and Clinicians (Experimental): Participants in this arm include children, adolescents, young adults (AYAs), caregivers, and clinicians. All participants will complete study-specific questionnaires at designated time points.
  Child/AYA/Caregiver Group: Participants will complete 3 questionnaires before the clinic visit and 2 questionnaires after the clinic visit.
  Clinician Group: Clinicians will complete 2 questionnaires after the clinic visit.
  Interventions: Behavioral: Age- and Role-Specific Questionnaire Administration

INTERVENTIONS:
Behavioral: Age- and Role-Specific Questionnaire Administration — Participants will be assigned a sequence number upon eligibility confirmation. The intervention consists of completing a series of questionnaires, as follows:
  Child/AYA/Caregiver Group:
  Pre-clinic Visit: 3 questionnaires (approximately 15-20 minutes total). Post-clinic Visit: 2 questionnaires (approximately 5-10 minutes total).
  Clinician Group:
  Post-clinic Visit: 2 questionnaires (approximately 5 minutes total).

SUMMARY:
The purpose of this project is to pilot test an electronically delivered symptom assessment tool Pediatric Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (Ped-PRO-CTCAE), completed by children/adolescents and young adults (AYAs) and caregivers and shared with their clinicians during an outpatient clinic visit, in preparation for a future test of intervention efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. First diagnosis of cancer
2. Receiving cancer therapy: surgery, myelosuppressive chemotherapy and/or radiation
3. 7-21 years of age
4. Completed at least 1 month of cancer chemotherapy treatment and are within 7-28 days of starting a treatment cycle or during ongoing therapy, followed at least every month in clinic
5. If surgery was part of treatment, the patient must be 3-6 weeks post surgery before participating in study
6. Caregiver must be present and 18 years and older.
7. Ability to understand and the willingness to personally sign the written IRB approved informed consent or assent document as appropriate.

Exclusion Criteria:

1. Child must be able to read or listen to and understand English and not have cognitive/memory impairments determined by the child's clinician
2. Caregiver must be able to read and understand English.

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Utilizing Ped-PRO-CTCAE for Clinician Access to Child/AYA and Caregiver Proxy Symptom Reports During Clinic Visits | 1 year
  To determine the feasibility of providing clinicians with child/AYA and caregiver (proxy) subjective symptom reports using the validated Ped-PRO-CTCAE items during a clinic visit.
Evaluation of Usability and Acceptability of Child/Adolescent and Caregiver Symptom Reports (Ped-PRO-CTCAE) for Clinicians in an Outpatient Oncology Clinic Setting | 1 year
  To evaluate the usability and acceptability of providing the child/adolescent and caregiver symptom reports (Ped-PRO-CTCAE) to the clinician in an outpatient oncology clinic setting
Analysis of Symptom-Related Outcome Variables to Inform Sample Size Calculations for a Future Randomized Clinical Trial of the Ped-PRO-CTCAE Intervention | 1 year
  To describe and analyze symptom-related outcome variables that will assist in sample size calculations for a future randomized clinical trial of the Ped-PRO-CTCAE intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Pyke-Grimm, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States